CLINICAL TRIAL: NCT03174249
Title: Leaving the Wheelchair Behind - Treating CRPS-II With Exposure Therapy Combined With Cortical Interventions: a Series of Case Reports
Brief Title: Exposure Therapy Combined With Cortical Interventions for CRPS-II
Acronym: ETHICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Folksam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FF-S23
Record Dates: First submitted 2017-03-28; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Behavioural therapy; Exposure in vivo; Cortical reorganisation; Mirror therapy
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Implosive Therapy; Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: A series of case-studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure therapy (Experimental): Graded exposure therapy in vivo in combination with methods targeting cortical reorganisation.
  Interventions: Behavioral: Exposure therapy

INTERVENTIONS:
Behavioral: Exposure therapy — Daily training at an in-patient ward during four plus four weeks, separated by a home training period of 6-8 weeks.
  Other Names: Mirror therapy; Desensibilisation training; Sensory re-education

SUMMARY:
Consecutive patients with long-standing complex regional pain syndrome II in a lower limb are treated with graded exposure therapy in vivo in combination with methods targeting cortical reorganisation.

DETAILED DESCRIPTION:
Complex regional pain syndrome, CRPS, is an uncommon but often very handicapping chronic pain syndrome. Most often, a single extremity is affected. The diagnosis is subdivided in CRPS type I where no nerve injury has been identified, and CRPS type II when a major nerve injury has been verified. With the exception of spontaneous pain, several of the symptoms related to CRPS may be connected to the inactivity and immobilization often seen in the history of CRPS patients.

Exposure in vivo, a form of behaviour therapy where the patient is gradually confronted with the avoided movements and activities, has been shown safe and effective for patients with CRPS type I. The present study uses a combination of exposure in vivo and interventions targeting a supposed cortical reorganisation with the hypothesis that the functional impairments would decrease, independent of possible changes in pain levels.

Consecutive patients with long-standing CRPS-II, diagnosed according to the Budapest criteria, in a lower limb are included. Treatment comprises daily graded exposure therapy in vivo, in combination with methods targeting cortical reorganisation: mirror therapy, desensibilisation training, and sensory re-education. The treatment is implemented at an in-patient ward during four plus four weeks, separated by a home training period of 6-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Complex regional pain syndrome II

Exclusion Criteria:

* Severe psychiatric disorder drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Photograph series of daily activities, PHODA | 12 weeks
  A measure of avoidance of activities - the subject reports level of hesitation in performing a number of everyday activities on a 0-100 rating scale.

SECONDARY OUTCOMES:
The Tampa Scale of Kinesiophobia - Short Form, TSK-SF | 12 weeks
  Fear of movement, assessed with a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Gordh, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala university hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No